CLINICAL TRIAL: NCT00792103
Title: An Open-Label Study to Evaluate the Safety of NP101, a Sumatriptan Iontophoretic Transdermal Patch, in the Treatment of Acute Migraine Over 12 Months
Brief Title: An Open-Label Study to Evaluate the Safety of NP101 in the Treatment of Acute Migraine Over 12 Months
Acronym: NP101-008
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROT-15-NP101-008
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NP101 (Experimental): sumatriptan iontophoretic transdermal patch
  Interventions: Drug: NP101

INTERVENTIONS:
Drug: NP101 — NP101 study patch 4 hour application

SUMMARY:
The primary objective is to evaluate the safety of long-term treatment with NP101 as assessed by:

* Subject self-examination skin irritation scores
* Adverse events
* Changes in vital signs and ECG parameters

The secondary objective is to evaluate the long term efficacy of NP101 as assessed by:

* Headache pain free at two hours after patch activation for all initial acute migraine attacks treated with NP101
* Headache pain relief at two hours after patch activation for all initial acute migraine attacks treated with NP101
* Nausea free at two hours after patch activation for all initial acute migraine attacks treated with NP101
* Phonophobia free at two hours after patch activation for all initial acute migraine attacks treated with NP101
* Photophobia free at two hours after patch activation for all initial acute migraine attacks treated with NP101
* Migraine free at two hours after patch activation for all initial acute migraine attacks treated with NP101

This study will use an open-label design to assess the long term safety of NP101 (sumatriptan iontophoretic transdermal patch).

Subjects who continue to be in good health (use of a triptan or use of an NP101 patch is not contraindicated) and received treatment (patch activation) with the study patch for a qualifying migraine under study NP101-007 will be considered eligible for enrollment into the open-label study. Subjects will be expected to remain in the study for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously enrolled in study NP101-007 and treated (patch activation) a qualifying migraine.
* Subject will be judged to be in good health, based upon the results of a medical history, physical examination, vital signs, and ECG. Subjects will not have any clinically significant abnormal vital signs or ECG parameters in order to qualify for enrollment. ECG must be done at enrollment for NP101-008 unless ECG for the Final Visit of study NP101-007 was conducted within 30 days.
* Female subjects of childbearing potential (not surgically sterile or 2 years post menopausal) must have a negative pregnancy test at enrollment.

Exclusion Criteria:

* Subject has less than two potential skin application sites.
* Subject has clinically significant abnormal vital signs or ECG parameters or had an adverse event while participating in NP101-007 that would preclude the continued treatment with the NP101 patch.
* Subject has had changes in their medical history or medication use that would preclude their use of sumatriptan as per the approved Imitrex® product Prescribing Information (PI) or their safe use of NP101 as per the NP101 Investigator's Brochure.
* Subject has or plans to start, stop, change treatment or dose of any of the following within 3 months prior to the subject's study Enrollment date and through the Final Visit: anxiolytics, lithium and other mood stabilizers such as valproate, carbamazepine or lamotrigine, hypnotics or antipsychotics.
* Subject has taken non-triptan serotonergic drugs including selective serotonin reuptake inhibitor (SSRI), serotonin and norepinephrine reuptake inhibitor (SNRI), tricyclic antidepressants (TCAs), monoamine oxidase inhibitor (MAOI) or preparations containing St. John's Wort within 1 month prior to enrollment and/or is planning to start any of these medications during the study (through Final Visit).
* Female subjects who are pregnant, breast feeding, or of childbearing potential, and are not using or are unwilling to use an effective form of contraception during the study and for a period of 30 days following Final Visit. Acceptable methods of contraception include barrier method with spermicide, intrauterine device (IUD), steroidal contraceptive (oral, transdermal, implanted or injected) or abstinence. If the exclusive male partner is surgically sterile, this will be acceptable.
* Subject has participated in a clinical study within 30 days of enrollment (excluding NP101-007) or is planning to participate in another clinical study for the duration of NP101-008.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pierce, MD PhD, Study Chair — NuPathe Inc.
Locations (34):
- United States (34):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Newport Beach, California
  - San Francisco, California
  - Santa Monica, California
  - Fairfield, Connecticut
  - Ocala, Florida
  - Palm Beach Gardens, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Decatur, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Springfield, Missouri
  - St Louis, Missouri
  - Mount Vernon, New York
  - Plainview, New York
  - Greensboro, North Carolina
  - West Chester, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wynnewood, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington

REFERENCES:
- [Derived] Smith TR, Goldstein J, Singer R, Pugach N, Silberstein S, Pierce MW. Twelve-month tolerability and efficacy study of NP101, the sumatriptan iontophoretic transdermal system. Headache. 2012 Apr;52(4):612-24. doi: 10.1111/j.1526-4610.2012.02094.x. Epub 2012 Feb 21. PMID 22352764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated January 2009 and completed in September 2010. Patients were enrolled from 34 investigative sites across the United States.
Pre-assignment Details: This was an open-label study to assess the long-term safety of NP101. Subjects who continued to be in good health and received treatment with an NP101 patch for a qualifying migraine in the pivotal NP101-007 study were considered eligible for enrollment.
Groups:
- NP101: The NP101 patch contained 86 mg of sumatriptan and was designed to deliver approximately 6.5 mg of sumatriptan over 4 hours. Patients were asked to use study patches to treat migraine episodes with moderate or severe headache pain for up to 12 months, during which they were permitted to apply (to the upper arms or thighs) a maximum of 6 patches within a 30-day period.
Period: Overall Study
Arm/Group | NP101
Started | 198 (15 subjects were enrolled but did not treat for a total of 183 subjects in the safety population)
Completed | 65
Not Completed | 133
Not completed — Enrolled, not treated | 15
Not completed — Lost to Follow-up | 17
Not completed — Adverse Event | 25
Not completed — Withdrawal by Subject | 52
Not completed — Protocol Violation | 10
Not completed — Did not apply 6 patches in 1st 3 mths | 14

BASELINE CHARACTERISTICS:
Population: Per protocol, the intent-to-treat (ITT) population was defined as all subjects who applied and activated at least one NP101 study patch and had at least one post baseline assessment for each migraine symptom (pain, photophobia, phonophobia, and nausea). Of the 183 subjects who applied at least one study patch, 181 subjects met the ITT criteria.
Arm/Group | NP101
Number analyzed (Participants) | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 183
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 183

OUTCOME MEASURES:

1. Secondary Outcome: Pain Relief
Description: Headache pain relief (no pain or mild headache pain) at two hours post activation of NP101.
Time Frame: 2 hours
Population: Per protocol, the intent-to-treat population was defined as all subjects who applied and activated at least one NP101 study patch and had at least one post baseline assessment for each migraine symptom (pain, photophobia, phonophobia, and nausea). Two treated subjects in the safety population did not meet this criteria.
Measure: Number; unit: participants
Arm/Group | NP101
Number analyzed (Participants) | 181
participants | 105 (0.341)

2. Primary Outcome: Subject Self-examination of Skin Irritation
Description: For each patch application, subjects performed a self-examination of skin irritation using a 5-point scale (0=no redness; 1=minimal skin redness; 2=moderate skin redness with sharp borders; 3=intense skin redness with or without swelling; 4=intense skin redness with blisters or broken skin).
Time Frame: 24 hours post patch activation
Population: Per protocol, the intent-to-treat population was defined as all subjects who applied and activated at least one NP101 study patch and had at least one post baseline assessment for each migraine symptom (pain, photophobia, phonophobia, and nausea).
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: NP101 Patches
Arm/Group | NP101
Number analyzed (Participants) | 183
Number analyzed (NP101 Patches) | 1917
scores on a scale | 1.0 (0.96)

3. Secondary Outcome: Nausea Free
Description: Nausea free at two hours after patch activation.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NP101
Number analyzed (Participants) | 181
participants | 143

4. Secondary Outcome: Phonophobia Free
Description: Phonophobia free at two hours after patch activation.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NP101
Number analyzed (Participants) | 181
participants | 109

5. Secondary Outcome: Photophobia Free
Description: Photophobia free at two hours after patch activation.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | NP101
Number analyzed (Participants) | 181
participant | 97

ADVERSE EVENTS:
Time Frame: All adverse events were collected from study enrollment until 30 days after the last patch application.
Arm/Group | NP101
Serious Adverse Events (participants affected / at risk) | 2/183
Other Adverse Events (participants affected / at risk) | 66/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NP101 (N=183)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NP101 (N=183)
Application site hypersensitivity (General disorders) | 11 (11)
Application Site Pain (General disorders) | 39 (39)
Application site pruritus (General disorders) | 40 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the study agreement, Investigators have the right to publish or present information and/or data arising from the study, provided the text of any such publication or presentation is submitted for review at least thirty days prior to submission for publication or other disclosure and NuPathe shall have the right to request the removal of any confidential information.